CLINICAL TRIAL: NCT00830986
Title: Cognition Following Computer Assisted Total Knee Arthroplasty: A Prospective Cohort Study
Brief Title: Cognition Following Computer Assisted Total Knee Arthroplasty
Acronym: Minimental
Status: Completed | Type: Observational
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Javad Parvizi, Rothman Institute of Orthopaedics
Other Study IDs: RIUWHOZ 09-01
Record Dates: First submitted 2009-01-26; First posted 2009-01-28 (Estimated); Last update posted 2009-04-16 (Estimated); Status verified 2009-01

CONDITIONS: Cognition; Embolism, Fat
Keywords: Mental Cognition Change; Fat Embolism; Bone Marrow Debris Emboli; Computer Assisted Total Knee Arthroplasty; Conventional Instrumented Total Knee Arthroplasty
MeSH Terms: conditions — Embolism, Fat | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Computer Assisted Total Knee Arthroplasty
  Interventions: Device: Total Knee Arthroplasty Implant (Scorpio®)
- 2: Conventional Instrumented Total Knee Arthroplasty
  Interventions: Device: Total Knee Arthroplasty Implant (Scorpio®)

INTERVENTIONS:
Device: Total Knee Arthroplasty Implant (Scorpio®) — Implantation of a Total Knee Arthroplasty using Conventional Intramedullary Instrumentation
  Other Names: Scorpio Total Knee Arthroplasty
  Groups: 2
Device: Total Knee Arthroplasty Implant (Scorpio®) — Implantation of a Total Knee Arthroplasty using a Computer Assisted Software, without Intramedullary Instrumentation
  Other Names: Scorpio Total Knee Arthroplasty
  Groups: 1

SUMMARY:
A significant number of patients experience postoperative cognitive changes following total joint arthroplasty. Among other causes, the mental status change may be the result of fat and bone marrow debris embolization. We hypothesized that the use of computer assisted total knee arthroplasty, which does not utilize intramedullary alignment rods, would produce less fat and bone marrow debris embolization and, hence, fewer mental status changes.

DETAILED DESCRIPTION:
Inclusion criteria

* Primary, cemented knee arthroplasty
* Unilateral or bilateral TKA

Exclusion criteria

* Patient is unable to speak English
* Unable to read and write
* Patient with history of psychiatric disorders (Depression, Schizophrenia, anxiety, bipolar dis.)
* Patients with history of IV drug abuse
* Previous history of dementia
* Patients on mental status changing medications

ELIGIBILITY:
Inclusion Criteria:

* Primary, cemented knee arthroplasty
* Unilateral or bilateral TKA

Exclusion Criteria:

* Patient is unable to speak English
* Unable to read and write
* Patient with history of psychiatric disorders (Depression, Schizophrenia, anxiety, bipolar dis.)
* Patients with history of IV drug abuse
* Previous history of dementia
* Patients on mental status changing medications

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 100 Consecutive patients requiring a total knee arthroplasty for degenerative arthritis of the knee
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2005-07; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Folstein Mini Mental State Examination (MMSE) | 6 Months Post-Operative

CONTACTS AND LOCATIONS:
Overall Officials: Javad Parvizi, MD, FRCS, Principal Investigator — Rothman Institute of Orthopaedics